CLINICAL TRIAL: NCT05408117
Title: Impact of Suture Type on Pigment Disturbances in Patients of Skin of Color: A Prospective, Randomized Split-wound Study
Brief Title: Impact of Suture Type on Pigment Disturbances in Patients of Skin of Color
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melissa Pugliano-Mauro (Other)
Responsible Party: Sponsor-Investigator, Melissa Pugliano-Mauro, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY22020176
Record Dates: First submitted 2022-05-30; First posted 2022-06-07 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Scar
Keywords: skin of color; split-wound; polypropylene; fast gut; pigmentary disturbance
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: prospective, randomized split-wound study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Sutures will be removed in their entirety before scar assessment by a co-investigator such that the outcomes assessor is blinded to which suture was used on which side of the scar.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- A= left/superior half of wound (Experimental): Patients with skin of color undergoing dermatologic surgery with planned standard elliptical excision with wound length of 3 cm or greater
  Interventions: Device: 5-0 Polypropylene epidermal suture; Device: 5-0 Fast gut epidermal suture
- B= right/inferior half of wound (Experimental): Patients with skin of color undergoing dermatologic surgery with planned standard elliptical excision with wound length of 3 cm or greater
  Interventions: Device: 5-0 Polypropylene epidermal suture; Device: 5-0 Fast gut epidermal suture

INTERVENTIONS:
Device: 5-0 Polypropylene epidermal suture — Split-wound, intra-individual comparison - half of wound will receive 5-0 polypropylene epidermal suture and half of wound will receive 5-0 fast gut epidermal suture
Device: 5-0 Fast gut epidermal suture — Split-wound, intra-individual comparison - half of wound will receive 5-0 polypropylene epidermal suture and half of wound will receive 5-0 fast gut epidermal suture

SUMMARY:
The present study assesses if dissolvable (fast gut) or non-dissolvable (polypropylene) epidermal sutures produce better cosmetic results in terms of dyspigmentation and scarring in patients of skin of color. Through a split-wound study design, patients undergoing standard elliptical excisions at least 3 cm in length will receive each suture type. Measurements of dyspigmentation and scarring will be made at 7 days (for the head and neck), 10 days (for the trunk and extremities), and 3 months for all locations.

DETAILED DESCRIPTION:
Subjects who consent to the study will have the following information recorded on the date of surgery: age, sex, indication for surgery, surgical site, scar length, size and type of buried intradermal suture, experience of surgeon (attending, fellow or resident), and New Immigration Scale (NIS) skin color. Basic patient medical data pertinent to wound healing/scar formation will be extracted from the medical record including history of hypertrophic scar/keloids, smoking, diabetes mellitus, and immunosuppression.

The subjects will undergo elliptical excision per standard of care. A single polyglactin 910 suture buried intradermal suture will be placed at the center of the wound. If additional buried intradermal sutures are needed, they will be placed equidistant from the center of the wound such that each side has an equivalent number of intradermal sutures. 5-0 polyglactin 910 will be used for wounds on the head and neck and 3-0 or 4-0 polyglactin 910 will be used for wounds on the trunk and extremities.

Following placement of the intradermal sutures, the subject's wound will be demarcated into halves, labeled either "A" or "B." "A" refers to the left or the superior side, and "B" refers to the right or inferior side. Prior to the study commencement, "A=fast gut" will be written on 17 index cards and "B=fast gut" will be written on 17 index cards. The index cards will be sealed in individual envelopes, shuffled to randomize, and stored securely with the study materials. At the time of surgery, the surgeon will randomly select an envelope which indicates which side will receive which suture type (either 5-0 fast absorbing gut or 5-0 polypropylene). This size of epidermal sutures will be used regardless of site of wound. The intervention will be applied sequentially with side A always being closed first. A simple running suture will be used on each half. The surgeon will aim to keep suture technique including spacing and distance from wound edge identical.

Following the procedure, a standard dressing will be applied and wound care will be discussed. Patients will be seen, as is routinely performed clinically, for suture removal for the polypropylene side in 7 days if the closure was on the head and neck and 10 days if the closure was on the trunk or extremities. Any residual component of fast gut suture that has not yet dissolved will be removed by the medical assistant or nurse so that the physician observer is blinded to which sutures were placed on which side. The following information will be collected at this suture removal visit:

* Photo of the scar
* Patients will perform the patient portion of the POSAS (Patient and Observer Scar Assessment Scale), a validated scale of scar cosmesis.
* A co-investigator not present at the time of the surgical procedure will perform the physician portion of the POSAS
* Scar width will be measured 1 cm from midline on each side of the wound. Measurements will be recorded in 0.5 mm increments.
* Pain incurred with suture removal will be measured via a 10 point Visual Analog Scale immediately after sutures are removed, with 1 representing no pain and 10, the worst pain imaginable.

Patients will be asked to return for an in person clinic visit 3 months after surgery for subsequent scar assessment. All surgical patients, not just those involved in the research study, have follow up appointments for suture removal at 7-14 days and at 3-6 months, as per physician discretion. This time interval is the standard of care. The following information will be collected at 3 month follow up:

* Photo of the scar
* Patient and observer POSAS scores (again, a co-investigator not present at the time of the surgical procedure will perform the physician portion of the POSAS).
* Dermatoscopic images of each side of the scar and of an area of normal skin. The dermatoscopic images will be used to calculate a skin hyperpigmentation index (SHI) score, a validated objective measure of skin hyperpigmentation (https://shi.skinimageanalysis.com).
* Scar width will be measured 1 cm from midline on each side of the wound. Measurements will be recorded in 0.5 mm increments.
* Clinical evidence of surgical site infection, wound disruption, and/or any other postsurgical complications.

Patients who fail to attend the in-person 3 month follow up visit will be contacted by telephone to complete the patient portion of the POSAS and asked to upload photos of the scar to their medical record via MyUPMC. Storage of images of the scars will occur for all patients, not just those participating in the study.

Upon completion of study visits, POSAS, SHI and other clinical data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Undergoing dermatologic surgery with planned standard elliptical excision with wound length of 3 cm or greater. Benign and malignant lesions will be included, including those that have undergone Mohs micrographic surgery prior to standard linear closure. All body sites will be included.
3. Able to give informed consent
4. Able to return for 3 month follow up
5. New Immigration Scale (NIS) skin color 4 or greater - The NIS is an 11 point scale, ranging from zero to 10, with zero representing albinism and 10 representing the darkest possible skin.

Exclusion Criteria:

1. High-tension closures not amenable to 5-0 simple running epidermal sutures
2. Known allergy to suture material
3. Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
POSAS | Suture removal date which is 7 days from the procedure if the excision is on the head or neck and 10 days from the procedure if the excision is on the trunk or extremities
  Patient and Observer Scar Assessment Scale (POSAS) outcome (6-60 scale). 6 subscales (which assess scar pain, itch, color, stiffness, thickness, and irregularity) comprise the POSAS measure and each are measured 1-10. Subscales will be summed to get a total score out of 60. Higher values represent worse outcomes.
POSAS | 3 months from procedure
  Patient and Observer Scar Assessment Scale (POSAS) outcome (6-60 scale). 6 subscales (which assess scar pain, itch, color, stiffness, thickness, and irregularity) comprise the POSAS measure and each are measured 1-10. Subscales will be summed to get a total score out of 60. Higher values represent worse outcomes.
Skin hyperpigmentation index | 3 months from procedure
  1-4 scale, higher value indicates worse outcomes (greater dyspigmentation), lower values represent better outcomes

SECONDARY OUTCOMES:
Scar width | Suture removal date which is 7 days from the procedure if the excision is on the head or neck and 10 days from the procedure if the excision is on the trunk or extremities
  Using a ruler to measure scar width 1 cm from midline on each side of the wound. Measurements will be recorded in 0.5 mm increments.
Scar width | 3 months from procedure
  Using a ruler to measure scar width 1 cm from midline on each side of the wound. Measurements will be recorded in 0.5 mm increments.
Complications | Suture removal date which is 7 days from the procedure if the excision is on the head or neck and 10 days from the procedure if the excision is on the trunk or extremities
  Incidence of surgical site infection, wound dehiscence, keloids, hematomas, suture abscesses, seromas, necrosis, and suture granulomas. Greater incidence represents worse outcomes.
Complications | 3 months from procedure
  Incidence of surgical site infection, wound dehiscence, keloids, hematomas, suture abscesses, seromas, necrosis, and suture granulomas. Greater incidence represents worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Pugliano-Mauro, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (3):
- United States (3):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Shadyside Place, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrne M, Aly A. The Surgical Suture. Aesthet Surg J. 2019 Mar 14;39(Suppl_2):S67-S72. doi: 10.1093/asj/sjz036. PMID 30869751
- [Background] Eisen DB, Zhuang AR, Hasan A, Sharon VR, Bang H, Crispin MK. 5-0 Polypropylene versus 5-0 fast absorbing plain gut for cutaneous wound closure: a randomized evaluator blind trial. Arch Dermatol Res. 2020 Apr;312(3):179-185. doi: 10.1007/s00403-019-02009-5. Epub 2019 Nov 13. PMID 31724097
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Tuinebreijer WE, Middelkoop E, Kreis RW, van Zuijlen PP. The patient and observer scar assessment scale: a reliable and feasible tool for scar evaluation. Plast Reconstr Surg. 2004 Jun;113(7):1960-5; discussion 1966-7. doi: 10.1097/01.prs.0000122207.28773.56. PMID 15253184
- [Background] Sklar LR, Pourang A, Armstrong AW, Dhaliwal SK, Sivamani RK, Eisen DB. Comparison of Running Cutaneous Suture Spacing During Linear Wound Closures and the Effect on Wound Cosmesis of the Face and Neck: A Randomized Clinical Trial. JAMA Dermatol. 2019 Mar 1;155(3):321-326. doi: 10.1001/jamadermatol.2018.5057. PMID 30649154
- [Background] Eilers S, Bach DQ, Gaber R, Blatt H, Guevara Y, Nitsche K, Kundu RV, Robinson JK. Accuracy of self-report in assessing Fitzpatrick skin phototypes I through VI. JAMA Dermatol. 2013 Nov;149(11):1289-94. doi: 10.1001/jamadermatol.2013.6101. PMID 24048361